CLINICAL TRIAL: NCT04167644
Title: Proper Timing of Control of Hypertension and Outcome in Acute Spontaneous Intracerebral Hemorrhage.
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital 7
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Intra Cerebral Hemorrhage; Hypertension
Keywords: ICH, Hypertension, GCS , and mRS.
MeSH Terms: conditions — Cerebral Hemorrhage; Hypertension; Hepatitis, Infectious Canine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unfavorable outcome: 80 patients with poor outcome were classified according to mRS score after discharge (mRS range from 3 up to 6).
  Interventions: Diagnostic Test: Modified Rankin Scale (mRS)
- Favorable outcome: 70 patients with better outcome were classified according to mRS score after discharge (mRS range from 0 up to 2) .
  Interventions: Diagnostic Test: Modified Rankin Scale (mRS)

INTERVENTIONS:
Diagnostic Test: Modified Rankin Scale (mRS) — Modified Rankin Scale (mRS) is a profoundly valid and reliable measure of disability and is broadly utilized for assessing stroke outcomes and degree of disability. We characterized a favorable outcome as mRS ranging from zero up to two, while unfavorable outcome ranging for 3 up to six

SUMMARY:
The ideal management of blood pressure in BP after acute intracerebral haemorrhage is still debated and whether a higher intensive reduction of blood pressure after acute intracerebral haemorrhage may be better or not is still controversial. Conflicting results from different randomized trials in regards to the clinical guidelines for management of hypertension in people with acute intracerebral hemorrhage (ICH). These results indicate that the management of BP and the prognosis after acute spontaneous ICH are very complicated.

Therefore, analysis based on actual blood pressure (BP) accomplished may be a more efficient method to assess the impact of BP management on outcome of ICH.

In our research, blood pressure (BP) management and prognosis were studied in patients with acute intracerebral hemorrhage to decide the perfect time control BP to improve outcome.

DETAILED DESCRIPTION:
Methods:

Patients were diagnosed by clinical examination and according to the initial CT brain after the onset of ICH.

Intensive management of blood pressure (BP) started once the diagnosis of intracerebral hemorrhage was established. Systolic blood pressure targeted 140 mm Hg by IV drug that lower BP like nicardipine or diltiazem. Oral antihypertensive medications like (Angiotensin II Receptor Blockers (ARBs) or Ca-blocker), after 24 h of hospitalization, was utilized in combination and step by step changed from intravenous administration.

Patients were exposed to:

A) Complete history taking and complete clinical assessment including neurological and general examinations.

B) Initial Glasgow Coma Scale score at admission to hospital and patients according to GCS score were classified to 3 groups I (13-15), II (5-12), and III (3-4 ) according to Hemphill et al 2001.

C-Modified Rankin Scale (mRS) is a profoundly valid and reliable measure of disability and is broadly utilized for assessing stroke outcomes and degree of disability. We characterized a favorable outcome as mRS ranging from zero up to two, while unfavorable outcome ranging for 3 up to six].

D- Routine laboratory examinations including CBC, blood sugar, coagulation tests, renal and hepatic functions.

E- CT brain was accomplished for all patients at onset of admission to hospital to decide the characters of spontaneous intracerebral hemorrhage (ICH). The volume of the intracerebral hemorrhage was determined utilizing the ABC/2 method (A is the most great diameter on the most large ICH cut, B is the diameter perpendicular to A, while, C is the number of axial cuts of ICH multiplied by the thickness of cuts. Additionally, the location ICH (regardless of whether infra or supatrentorial), and if there is IVH or not, also, if there is shift of midline structure or hydrocephalic changes were determined. Regarding ICH volume, patients were partitioned into two groups (< 30 cm3 and ≥30 cm3).

Statistical analysis

SPSS version 19.0 was utilized for statistical analysis. Data were collected and displayed as numbers proportions, mean ± standard deviation, and range. Favorable and unfavorable groups were compared by chi-square measurement. For variable with ordinary distributions and homogeneous variances, Student's t-test was utilized to check the significant difference between the mean ± standard deviation values in the two groups. P value <0.05 were considered of statistical significant results.

Multivariate logistic regression analysis was accomplished for the independent variables or factors that were accompanied by better outcomes: like younger ages, GCS at admission, diastolic blood pressure one hour after admission, systolic BP 6 h after admission, and systolic blood pressure 24 h after admission.

ELIGIBILITY:
Inclusion Criteria:

- Patients incorporated into this study aged over 25 years of either sex with first spontaneous intracerebral hemorrhage (ICH).

Exclusion Criteria:

* Secondary ICH were excluded from this study (like traumatic, hemorrhagic infarcts, AVM, bleeding tumors or SOL, or IVH only without ICH).
* Patients with previous ischemic stroke or T1As

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study was conducted during the period from May 2018 to the end of April 2019. This study was conducted on150 patients presented by acute spontaneous intracerebral hemorrhage (ICH) were admitted to the Department of Neurology of Mansoura University Hospital. Modified Rankin Scale score (mRS) after discharge was calculated and accordingly, patients were partitioned into two main groups: The first group was favorable outcome patients (mRS queal 0-2) and the second group was unfavorable outcome patients (mRS queal 3-6). Independent factors that were significantly related to prognosis were assessed by multivariate logistic regression.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Glasgow Coma Scale score | 24 hours
  Initial Glasgow Coma Scale score at admission to hospital and patients according to GCS score were classified to 3 groups I (13-15), II (5-12), and III (3-4 ) according to Hemphill et al 2001.
CT brain | 24 hours
  CT brain was accomplished for all patients at onset of admission to hospital to decide the characters of spontaneous intracerebral hemorrhage (ICH). The volume of the intracerebral hemorrhage was determined utilizing the ABC/2 method (A is the most great diameter on the most large ICH cut, B is the diameter perpendicular to A, while, C is the number of axial cuts of ICH multiplied by the thickness of cuts. Additionally, the location ICH (regardless of whether infra or supatrentorial), and if there is IVH or not, also, if there is shift of midline structure or hydrocephalic changes were determined. Regarding ICH volume, patients were partitioned into two groups (< 30 cm3 and ≥30 cm3)

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 24 hours
  Modified Rankin Scale (mRS) is a profoundly valid and reliable measure of disability and is broadly utilized for assessing stroke outcomes and degree of disability. We characterized a favorable outcome as mRS ranging fModified Rankin Scale (mRS) is a profoundly valid and reliable measure of disability and is broadly utilized for assessing stroke outcomes and degree of disability. We characterized a favorable outcome as mRS ranging from zero up to two, while unfavorable outcome ranging for 3 up to six rom zero up to two, while unfavorable outcome ranging for 3 up to six

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Mufti F, Thabet AM, Singh T, El-Ghanem M, Amuluru K, Gandhi CD. Clinical and Radiographic Predictors of Intracerebral Hemorrhage Outcome. Interv Neurol. 2018 Feb;7(1-2):118-136. doi: 10.1159/000484571. Epub 2018 Jan 12. PMID 29628951
- [Background] Lattanzi S, Silvestrini M. Blood pressure in acute intra-cerebral hemorrhage. Ann Transl Med. 2016 Aug;4(16):320. doi: 10.21037/atm.2016.08.04. No abstract available. PMID 27668240
- [Background] Sakamoto Y, Koga M, Toyoda K. Response to letter regarding article, "Systolic blood pressure after intravenous antihypertensive treatment and clinical outcomes in hyperacute intracerebral hemorrhage: the stroke acute management with urgent risk-factor assessment and improvement-intracerebral hemorrhage study". Stroke. 2013 Nov;44(11):e153. doi: 10.1161/STROKEAHA.113.002903. Epub 2013 Sep 17. No abstract available. PMID 24046009
- [Background] Rabinstein AA. Optimal Blood Pressure After Intracerebral Hemorrhage: Still a Moving Target. Stroke. 2018 Feb;49(2):275-276. doi: 10.1161/STROKEAHA.117.020058. Epub 2018 Jan 4. No abstract available. PMID 29301975
- [Background] Wang X, Arima H, Heeley E, Delcourt C, Huang Y, Wang J, Stapf C, Robinson T, Woodward M, Chalmers J, Anderson CS; INTERACT2 Investigators. Magnitude of blood pressure reduction and clinical outcomes in acute intracerebral hemorrhage: intensive blood pressure reduction in acute cerebral hemorrhage trial study. Hypertension. 2015 May;65(5):1026-32. doi: 10.1161/HYPERTENSIONAHA.114.05044. Epub 2015 Mar 23. PMID 25801872
- [Background] Wang X, Arima H, Al-Shahi Salman R, Woodward M, Heeley E, Stapf C, Lavados PM, Robinson T, Huang Y, Wang J, Delcourt C, Anderson CS. Rapid Blood Pressure Lowering According to Recovery at Different Time Intervals after Acute Intracerebral Hemorrhage: Pooled Analysis of the INTERACT Studies. Cerebrovasc Dis. 2015;39(3-4):242-8. doi: 10.1159/000381107. Epub 2015 Mar 25. PMID 25823544
- [Background] Anderson CS, Heeley E, Huang Y, Wang J, Stapf C, Delcourt C, Lindley R, Robinson T, Lavados P, Neal B, Hata J, Arima H, Parsons M, Li Y, Wang J, Heritier S, Li Q, Woodward M, Simes RJ, Davis SM, Chalmers J; INTERACT2 Investigators. Rapid blood-pressure lowering in patients with acute intracerebral hemorrhage. N Engl J Med. 2013 Jun 20;368(25):2355-65. doi: 10.1056/NEJMoa1214609. Epub 2013 May 29. PMID 23713578
- [Background] Qureshi AI, Palesch YY, Barsan WG, Hanley DF, Hsu CY, Martin RL, Moy CS, Silbergleit R, Steiner T, Suarez JI, Toyoda K, Wang Y, Yamamoto H, Yoon BW; ATACH-2 Trial Investigators and the Neurological Emergency Treatment Trials Network. Intensive Blood-Pressure Lowering in Patients with Acute Cerebral Hemorrhage. N Engl J Med. 2016 Sep 15;375(11):1033-43. doi: 10.1056/NEJMoa1603460. Epub 2016 Jun 8. PMID 27276234
- [Background] Lattanzi S, Silvestrini M. Optimal achieved blood pressure in acute intracerebral hemorrhage: INTERACT2. Neurology. 2015 Aug 11;85(6):557-8. doi: 10.1212/01.wnl.0000470918.40985.d0. No abstract available. PMID 26259858
- [Background] Moullaali TJ, Wang X, Woodhouse LJ, Law ZK, Delcourt C, Sprigg N, Krishnan K, Robinson TG, Wardlaw JM, Al-Shahi Salman R, Berge E, Sandset EC, Anderson CS, Bath PM; BASC Investigators. Lowering blood pressure after acute intracerebral haemorrhage: protocol for a systematic review and meta-analysis using individual patient data from randomised controlled trials participating in the Blood Pressure in Acute Stroke Collaboration (BASC). BMJ Open. 2019 Jul 16;9(7):e030121. doi: 10.1136/bmjopen-2019-030121. PMID 31315876
- [Background] Qureshi AI, Palesch YY, Foster LD, Barsan WG, Goldstein JN, Hanley DF, Hsu CY, Moy CS, Qureshi MH, Silbergleit R, Suarez JI, Toyoda K, Yamamoto H; ATACH 2 Trial Investigators. Blood Pressure-Attained Analysis of ATACH 2 Trial. Stroke. 2018 Jun;49(6):1412-1418. doi: 10.1161/STROKEAHA.117.019845. Epub 2018 May 22. PMID 29789395
- [Background] Hemphill JC 3rd, Bonovich DC, Besmertis L, Manley GT, Johnston SC. The ICH score: a simple, reliable grading scale for intracerebral hemorrhage. Stroke. 2001 Apr;32(4):891-7. doi: 10.1161/01.str.32.4.891. PMID 11283388
- [Background] Banks JL, Marotta CA. Outcomes validity and reliability of the modified Rankin scale: implications for stroke clinical trials: a literature review and synthesis. Stroke. 2007 Mar;38(3):1091-6. doi: 10.1161/01.STR.0000258355.23810.c6. Epub 2007 Feb 1. PMID 17272767
- [Background] Maeda AK, Aguiar LR, Martins C, Bichinho GL, Gariba MA. Hematoma volumes of spontaneous intracerebral hemorrhage: the ellipse (ABC/2) method yielded volumes smaller than those measured using the planimetric method. Arq Neuropsiquiatr. 2013 Aug;71(8):540-4. doi: 10.1590/0004-282X20130084. PMID 23982013
- [Background] Hu TT, Yan L, Yan PF, Wang X, Yue GF. Assessment of the ABC/2 Method of Epidural Hematoma Volume Measurement as Compared to Computer-Assisted Planimetric Analysis. Biol Res Nurs. 2016 Jan;18(1):5-11. doi: 10.1177/1099800415577634. Epub 2015 Mar 23. PMID 25802386
- [Background] Shi J, Cai Z, Han W, Dong B, Mao Y, Cao J, Wang S, Guan W. Stereotactic Catheter Drainage Versus Conventional Craniotomy for Severe Spontaneous Intracerebral Hemorrhage in the Basal Ganglia. Cell Transplant. 2019 Aug;28(8):1025-1032. doi: 10.1177/0963689719852302. Epub 2019 May 27. PMID 31129993
- [Background] Ahmed Esmael, Mohammed El Sherif and Mohamed Saad. Prediction of 30-days Mortality of Intracerebral Hemorrhage by a Powerful but Easy to Use Intracerebral Hemorrhage Score. 2016; 6 (2): 1-11.
- [Result] Cordonnier C, Demchuk A, Ziai W, Anderson CS. Intracerebral haemorrhage: current approaches to acute management. Lancet. 2018 Oct 6;392(10154):1257-1268. doi: 10.1016/S0140-6736(18)31878-6. PMID 30319113